CLINICAL TRIAL: NCT07025161
Title: Brief Behavioral Intervention for Pain (Shepherd's Hope)
Brief Title: Brief Mindfulness Intervention for Patients at a Free Acute Care Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00004916 Shepherd's Hope
Record Dates: First submitted 2025-04-23; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Coping Information (Active Comparator): Participants will be randomized to listen to a 4-minute audio recording providing common pain coping techniques (e.g., ice, rest, medication, surgery).
  Interventions: Behavioral: Pain Coping Information
- Mindful Pain Management (Experimental): Participants will be randomized to listen to a 4-minute audio recording consisting of a 1-minute introduction to mindfulness followed by a 1-minute and 30-second mindful breathing practice and a 1-minute and 30-second mindfulness of pain practice.
  Interventions: Behavioral: Mindful Pain Management

INTERVENTIONS:
Behavioral: Pain Coping Information — A 4-minute audio recording providing common pain coping techniques (e.g., ice, rest, medication, surgery).
  Arms: Pain Coping Information
Behavioral: Mindful Pain Management — A 4-minute audio recording consisting of a 1-minute introduction to mindfulness followed by a 1-minute and 30-second mindful breathing practice and a 1-minute and 30-second mindfulness of pain practice.
  Arms: Mindful Pain Management

SUMMARY:
This is a single-site, two-arm, parallel-group randomized clinical trial (RCT). The clinical effects of a 4-minute audio-recorded mindfulness intervention for 100 English-speaking patients and 100 Spanish-speaking patients at a free acute care clinic will be investigated relative to a 4-minute audio-recoding about pain psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Seeking treatment at the Shepherd's Hope Downtown Clinic

Exclusion Criteria:

* Cognitive impairment preventing completion of study procedures.
* Other unstable illness judged by medical staff to interfere with study involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-04-21 (Estimated); Study Completion 2026-04-21 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.
Change in Anxiety Numeric Rating Scale | Immediately before to after 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no anxiety and 10 representing severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd's Hope Downtown Clinic, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
All our data is aggregate and anonymous.